CLINICAL TRIAL: NCT03800927
Title: Multi Week Long-Duration Ultrasound for Knee Osteoarthritis
Brief Title: Long-Duration Ultrasound for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OA-04
Record Dates: First submitted 2018-12-15; First posted 2019-01-11 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Intervention Model Description: Participants will receive active and sham devices for the first 12-weeks. Responders to treatment will continue with 12 weeks of additional active treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Ultrasound Device (Placebo Comparator): No ultrasound treatment
  Interventions: Device: Long duration ultrasound
- Active Ultrasound Device (Active Comparator): Active treatment
  Interventions: Device: Long duration ultrasound

INTERVENTIONS:
Device: Long duration ultrasound — Low-intensity long duration ultrasound treatment

SUMMARY:
This study will measure the 24-week pain relief from long-duration ultrasound on the symptoms of knee arthritis pain.

ELIGIBILITY:
Inclusion Criteria:

* Are you between 18 and 80 years of age (inclusive)?
* Can you speak, read, and write in English?
* Do you have knee pain that has lasted at least 3 months?
* Are you willing and able to self-administer the ultrasound device daily within your place of residence or during normal daily activity?
* Are you willing to keep all pain medications stable and discuss with the investigator any needs to change medications during the study period? This may include drugs administered topically, orally, transdermally, or by injection.
* Are you willing to document usage of any medications during the study period?
* Do you agree to discontinue all other interventional treatment modalities on the lower back during the study? (e.g., transcutaneous electric nerve stimulation [TENS], electronic muscle stimulation, traditional ultrasound, massage therapy, chiropractic services)
* On a Numeric Rating Scale (NRS) of 0 (no pain) to 10 (pain as bad as you can imagine), how would you rate your average pain over the past week? Pain must be ≥4 for the subject to be enrolled in this study. This criterion will be assessed by self-report at Visit 1.

Exclusion Criteria:

* Have you participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening?
* Are you pregnant?
* Are you a prisoner?
* Are you non-ambulatory (unable to walk)?
* Do you have a pacemaker?
* Do you have a malignancy in the treatment area?
* Do you have an active infection, open sores, or wounds in the treatment area?
* Do you have impaired sensation in the treatment area, such as caused by chemotherapy or anesthesia?
* Do you have a known neuropathy (disease of the brain or spinal nerves)?
* Do you have a hereditary disposition (tendency) for excessive bleeding (hemorrhage)?
* Do you have peripheral artery disease?
* Does the subject display any condition which, in the judgment of the investigator, would make participation in the study unacceptable including, but not limited to, the subject's ability to understand and follow instructions?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Units on a Numeric Rating Scale (NRS) | Average of first week (start of study) to average measure at 24 weeks (end of study)
  NRS on the scale of 1 - 10, 1 being minimum and 10 being maximum, Change was calculate from base line

SECONDARY OUTCOMES:
Function | First week (start of study) to 24 weeks (end of study)
  WOMAC questionnaire will be utilized (Western Ontario and McMaster Universities Arthritis Index) at baseline and post-treatment to calculate the change in the scores. WOMAC was divided into 3 categories: pain, stiffness, function and total score. The pain category consists of five scores from 0-10, 0 is no pain 10 is worst pain possible for a range of 0 - 50 points. The stiffness category consists of two scores from 0-10, 0 is no stiffness 10 is worst stiffness possible for a range of 0 - 20 points. The function score consists of 17 scores from 0-10, 0 is normal function and 10 is severely limited function, for a range of 0 - 170 points. Categories were multiplied by 10 for analysis. Total score is the sum of pain, stiffness, and function scores (range of 0 - 2400)
Strengthen | First week (start of study) to 24 weeks (end of study)
  Strength measurement with force meter (Newtons)
Range of motion | First week (start of study) to 24 weeks (end of study)
  Range of Motion measurement with motion machine (Degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Ortiz, MPH, DO, Study Director — Medical Pain Consultants
Locations (2):
- United States (2):
  - Orthopedic Foundation, Stamford, Connecticut
  - Medical Pain Consultants, Dryden, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Class II Medical Device — https://www.samrecover.com